CLINICAL TRIAL: NCT05606640
Title: Gaining Insight Into the Complexity of Pain in Patients With Haemophilia
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Prof. dr. Mira Meeús, Professor Rehabilitation Sciences and Physiotherapy, Universiteit Antwerpen
Other Study IDs: PAINSTUDY_2019; 2019/28OCT/469 (Other: CEHF); B300201942304 (Other: Belgian registration number); 19/43/483 (Other: University Hospital Antwerp); EDGE000540 (Other: University Hospital Antwerp)
Record Dates: First submitted 2022-10-28; First posted 2022-11-07 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: Haemophilia; arthropathy; Pain; Biopsychosocial
MeSH Terms: conditions — Hemophilia A; Hemophilia B; Joint Diseases; Pain | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Haemophilia: Adult males with severe or moderate haemophilia A or B
  Interventions: Diagnostic Test: Biopsychological pain assessment

INTERVENTIONS:
Diagnostic Test: Biopsychological pain assessment — At baseline (T0) patients underwent the somatosensory pain assessment, joint structure and function assessment and filled in all questionnaires. During one month after baseline (T1) patients wore an activity tracker and filled in the Illness Perceptions Questionnaire and the International Physical Activity questionnaire. During one year after the baseline assessment (T2) patients filled in every month The Brief Pain Inventory, Illness Perceptions Questionnaire and the EQ-5D-5L quality of life questionnaire.
  Other Names: Pain-related questionnaires: Brief Pain Inventory, Douleur Neuropathique en 4 questions, Central Sensitization Inventory; Psychological questionnaires: Pain Catastrophizing Scale, Hospital Anxiety and Depression Scale, Fear Avoidance and Beliefs Questionnaire, The EuroQol-5 (EQ-5D-5L) quality of life questionnaire; Functional questionnaires: Haemophilia Activity List, International Physical Activity Questionnaire (IPAQ); Joint structure: Magnetic Reasoning Imaging (MRI) ankles & ultrasound evaluation of affected joints; Joint function: Hemophilia Joint Health Score (HJHS 2.1), Timed Up & Go, 2 minutes walking test, activity tracker; Somatosensory pain assessment: Quantitative Sensory testing protocol, Conditioned Pain Modulation protocol

SUMMARY:
Joint pain has been reported as a major problem in people with haemophilia (PwH). Therefore, haemophilia in adults seems clinically more related to a musculoskeletal disorder than a bleeding disorder, with many patients reporting a pain intensity exceeding 6/10 on a visual analogue scale. However, although the complexity of joint pain has been studied in chronic joint pain conditions such as low back pain, osteoarthritis or rheumatoid arthritis, until present only very limited research has been done on joint pain within PwH. Therefore, exploring the underlying mechanisms and the functional implications of this intense joint pain is urgently needed. As such, the main aim of the current prospective observational study is to gain more insights in joint pain in PwH enabling us to move towards adequate pain management in PwH.

DETAILED DESCRIPTION:
In this study, adult patients with moderate or severe Haemophilia from the Haemophilia Treatment Centers will be invited to participate in the study. Patients willing to participate will be asked to complete a battery of questionnaires in the week prior to the study. Patients will undergo a comprehensive baseline evaluation after their regular appointment with their treating hematologist.

During the baseline assessment, the structure of ankle and knee joints will be assessed, using respectively magnetic resonance imaging (MRI) and ultrasound evaluation. Besides, patients will be asked to perform some active movements to quantify the physical functions of the lower limb and will undergo an extensive pain assessment.

During one month following baseline assessment, patients will be closely monitored. They will be asked to fill in a diary linked to their usual logbook in which they indicate the minimal and maximal intensity of pain, location of pain, intake of regular or additional (in case of bleeding) clotting factors, intake of analgesics, occurrence and location of assumed bleeding. Patients will be asked to wear an activity tracker to register the number of steps during this month.The short version of the International Physical Activity Questionnaire (IPAQ) will be used to evaluate the self-reported estimation of weekly physical activity.

During the next 11 months, patients will be asked to fill in three online pain-related questionnaires: the Brief Pain Inventory, Brief Illness Perception Questionnaire and the EQ-5D-5L questionnaire once a month.

ELIGIBILITY:
Inclusion Criteria:

* adult (18-65y) patients with moderate (i.e. between 1 and 5 % normal Factor activity) or severe (less than 1% normal Factor activity) Haemophilia A (i.e. Factor VIII deficiency) or B (i.e. Factor IX deficiency)
* Dutch or French speaking
* Patients who provide their haemophilia treatment regimen to be stable (i.e. a regular treatment during the last 6 months, verified by the existing patients' logbook).

Exclusion Criteria:

* Patients suffering from known neuropathies with definite medical causes independent from the haemophilia (e.g. diabetes polyneuropathy)
* Patients with a haemarthrosis in the month preceding study participation will be excluded as well. In case of doubt, ultrasound will be used to check the presence of bleed in the joint.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult males with moderate or severe Haemophilia A or B will be recruited from the Haemophilia Treatment Centers in Antwerp (Antwerp University Hosptial) and Brussels (Cliniques universitaires Saint-Luc). Age-matched healthy control subjects will be recruited from family and acquintances of the researchers and hospital/university personnel.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Pain localisation | At baseline (T0)
  The body chart of the Brief Pain Inventory (BPI) was used to investigate painful body sites.
Pain localisation | At one year follow-up (T2)
  The body chart of the Brief Pain Inventory (BPI) was used to investigate painful body sites.
Pain severity | At baseline (T0)
  The BPI was used to evaluate the individual's pain experience within the last 24 hours by four items, resulting in a total pain severity score. Minimum score 0, maximum score 10. The higher te score, the higher the pain severity.
Pain severity | At one year follow-up (T2)
  The BPI was used to evaluate the individual's pain experience within the last 24 hours by four items, resulting in a total pain severity score. Minimum score 0, maximum score 10. The higher te score, the higher the pain severity.
Pain interference | At baseline (T0)
  The BPI was used to evaluate how much pain interferes with patient's daily activities. This was assessed by seven items, resulting in a total pain interference score. Minimum score 0, maximum score 10. The higher the score, the more pain interference.
Pain interference | At one year follow-up (T2)
  The BPI was used to evaluate how much pain interferes with patient's daily activities. This was assessed by seven items, resulting in a total pain interference score. Minimum score 0, maximum score 10. The higher the score, the more pain interference.
Signs of neuropathic pain | At baseline (T0)
  The Douleur Neuropathique en 4 questions (DN4) was applied as a screening tool for the presence of a neuropathic pain component. Minimum score 0, maximum score 10, a score of ≥4/10 was used as a cut-off.
Signs of central sensitization | At baseline (T0)
  The Central Sensitisation Inventory (CSI) part A was used to identify signs of central sensitization (CS) i.e. increased sensitivity of nociceptive neurons in the central nervous system.The presence of 25 pain-related psychological, cognitive and functional signs are scored from 0 (never) to 4 (always). A total score exceeding ≥40/100 indicated central sensitization.
Pain Catastrophizing | At baseline (T0)
  The Pain Catastrophizing Scale (PCS) asked participants to reflect on previous painful experiences and to rate their degree of catastrophic thinking in the content domains of rumination, magnification and helplessness. A score of 0 (not at all) to 4 (all the time) was indicated for each of the 13 items, resulting in a total score range of 0-52. Higher scores were associated with higher levels of pain catastrophizing.
Anxiety and Depression | At baseline (T0)
  The Hospital Anxiety and Depression Scale (HADS) was used to establish symptoms of anxiety and depression. This 14-item questionnaire consists of two subscales each including 7 items, the first to identify anxiety and the second depression. Individual items were scored from 0 to 3, resulting in a total range score of 0-21 for each subscale. A score of ≥8/21 was determined as a cut-off, indicating anxiety and depression.
Fear Avoidance and Beliefs | At baseline (T0)
  The fear avoidance and beliefs questionnaire (FABQ) will be used to assess fear avoidance behaviors. The first five items question physical activity, the other 11 activities work. A minimum score is 0, maximum 24. Higher scores indicate fear avoidance behaviors.
Life quality | At baseline (T0)
  The EQ-5D-5L was used to assess quality of life. From five items investigating the impact of their disease, a health utility score was calculated. Additionally, the questionnaire consists of a visual analogue scale (VAS) labelled from 0: "worst imaginable health state," to 100 "best imaginable health state" providing the EQ-VAS.
Life quality | At one year follow-up (T2)
  The EQ-5D-5L was used to assess quality of life. From five items investigating the impact of their disease, a health utility score was calculated. Additionally, the questionnaire consists of a visual analogue scale (VAS) labelled from 0: "worst imaginable health state," to 100 "best imaginable health state" providing the EQ-VAS.
Haemophilia Activity Limitations | At baseline (T0)
  The Haemophilia Activity List (HAL) was used to assess activity limitations and participation restrictions people with haemophilia suffer with. A sum score and component scores can be calculated, resulting in scores ranging from 0-100. Lower scores represent higher levels of participation restrictions.
Physical endurance ability | At baseline (T0)
  The 2 minutes walking test (2MWT) was used as a performance-based test to assess their functional activity. Subjects were asked to walk as far as possible for two minutes in a 30 meters flat corridor, resulting in the walking distance in meters.
Physical functioning | At baseline (T0)
  The Timed Up & Go (TUG) consists of asking the patient to sit on a standard armchair; stand up and walk 3 meters; turn around at the line and walk back to the chair and sit down at a normal pace.
Joint structure US | At baseline (T0)
  Ultrasound (US) examinations will be performed with a linear probe (3-13 MHz) Esaote, type MyLab Gamma, Genova, Italy).The Haemophilia Early Arthropathy Detection with Ultrasound (HEAD-US) scanning procedure and scoring method will be performed by one of our investigators. A score of 0/8 (normal bone 0/2, normal cartilage 0/4, absent hypertrophic synovium 0/2) is considered normal. A score above 1/8 is considered as abnormal.
Joint structure MRI | At baseline (T0)
  Magnetic Reasoning Imaging (MRI) of the ankles will be performed with a 3T-magnet (GE Signa Premier, GE Healthcare, Milwaukee, USA).Joint images will be classified with the international Prophylaxis Study Group (IPSG) scale. Joints will be classified as abnormal if talocrural joints or subtalar joints were positive at IPSG-score. Joints will be considered healthy if the total score was of 1/17.
Illness perceptions | At baseline (T0)
  The illness perceptions questionnaire (B-IPQ) includes nine items ranging from 0 (minimum) to 10 (maximum) and questions the perceptions related to the patients disease. No total score exists, as each item is scored individually. Higher scores indicate more negative or unhelpful illness perceptions. A change score between baseline (T0) and one year follow-up (T2) will be calculated.
Illness perceptions | At one year follow-up (T2)
  The illness perceptions questionnaire (B-IPQ) includes nine items ranging from 0 (minimum) to 10 (maximum) and questions the perceptions related to the patients disease. No total score exists, as each item is scored individually. Higher scores indicate more negative or unhelpful illness perceptions. A change score between baseline (T0) and one year follow-up (T2) will be calculated.
Physical activity | At baseline (T0)
  The International Physical Activity Scale (IPAQ) questions the hours of physical activity over the last week (Higher scores are higher levels of physical activity). Based on the patient's answers a MET-minute score is calculated (MET-minutes x weight in kilograms/60kilograms)
Physical activity | At one month follow-up (T1)
  The International Physical Activity Scale (IPAQ) questions the hours of physical activity over the last week. Based on the patient's answers a MET-minute score is calculated (MET-minutes x weight in kilograms/60kilograms)
Joint function | At baseline (T0)
  Joint function of the ankles, knees and ankles was assessed with the HJHS 2.1. Minimum score is 0, maximum, 20. The higher the score the more functional limitations. HJHS scores are considered positive when scores reach 1/20.
Warm and cold detection threshold | At baseline (T0)
  Thermal hyper or hypo esthesia were assessed with a thermode attached at the dominant wrist by use of a validated Quantitative Sensory testing protocol with the Medoc TSA-2 device.
Warm and cold pain thresholds | At baseline (T0)
  Thermal hyper or hypo algesia were assessed with a thermode attached at the dominant wrist by use of a validated Quantitative Sensory testing protocol with the Medoc TSA-2 device.
Mechanical pain thresholds | At baseline (T0)
  Mechanical local and widespread hyperalgesia indicated by lower pressure pain thresholds were assessed with a digital algometer at the knee joints, ankle joints and forehead. This by use of a validated quantitative sensory testing protocol.
Temporal summation of pain | At baseline (T0)
  Temporal summation (or bottom-up sensitization) of pain was assessed by use of a 60g Von Frey monofilament at the medial knee and dorsal side of the wrist of the dominant side.
Conditioned Pain Modulation | At baseline (T0)
  Dysfunctional endogenous pain inhibition (as form of central pain processing) was assessed by a validated protocol applying the Medoc TSA-2 device with thermodes attached at both wrists.

SECONDARY OUTCOMES:
Pain interference change | Change from baseline (T0) to one year follow-up (T2)
  The BPI was used to evaluate how much pain interferes with patient's daily activities. This was assessed by seven items, resulting in a total pain interference score. Minimum score 0, maximum score 10. The higher the score, the more pain interference.A change score between baseline and one year follow-up will be calculated.
Pain severity change | Change from baseline (T0) to one year follow-up (T2)
  The BPI was used to evaluate the individual's pain experience within the last 24 hours by four items, resulting in a total pain severity score. Minimum score 0, maximum score 10. The higher te score, the higher the pain severity.A change score between baseline (T0) and one year follow-up (T2) will be calculated.
Fear Avoidance and beliefs change | Change from baseline (T0) to one year follow-up (T2)
  The fear avoidance and beliefs questionnaire (FABQ) will be used to assess fear avoidance behaviors. The first five items question physical activity, the other 11 activities work. A minimum score is 0, maximum 24. Higher scores indicate fear avoidance behaviors. A change score between baseline (T0) and one year follow-up (T2) will be calculated.
Anxiety and Depression change | Change from baseline (T0) to one year follow-up (T2)
  The Hospital Anxiety and Depression Scale (HADS) was used to establish symptoms of anxiety and depression. This 14-item questionnaire consists of two subscales each including 7 items, the first to identify anxiety and the second depression. Individual items were scored from 0 to 3, resulting in a total range score of 0-21 for each subscale. A score of ≥8/21 was determined as a cut-off, indicating anxiety and depression.A change score between baseline (T0) and one year follow-up (T2) will be calculated.
Illness Perceptions change | Change from baseline (T0) to one year follow-up (T2)
  The illness perceptions questionnaire (B-IPQ) includes nine items ranging from 0 (minimum) to 10 (maximum) and questions the perceptions related to the patients disease. No total score exists, as each item is scored individually. Higher scores indicate more negative or unhelpful illness perceptions. A change score between baseline (T0) and one year follow-up (T2) will be calculated.
Pain Catastrophizing change | Change from baseline (T0) to one year follow-up (T2)
  The Pain Catastrophizing Scale (PCS) asked participants to reflect on previous painful experiences and to rate their degree of catastrophic thinking in the content domains of rumination, magnification and helplessness. A score of 0 (not at all) to 4 (all the time) was indicated for each of the 13 items, resulting in a total score range of 0-52. Higher scores were associated with higher levels of pain catastrophizing. A change score between baseline (T0) and one year follow-up (T2) will be calculated.
Pain localisation change | Change from baseline (T0) to one year follow-up (T2)
  The body chart of the Brief Pain Inventory was used to investigate painful body sites. A change score between baseline (T0) and one year follow-up (T2) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Roussel, Principal Investigator — Universiteit Antwerpen; Cedric Hermans, Principal Investigator — Cliniques universitaires Saint-Luc / UCLouvain; Catherine Lambert, Principal Investigator — Cliniques universitaires Saint-Luc / UCLouvain; Sébastien Lobet, Principal Investigator — Cliniques universitaires Saint-Luc / UCLouvain; Philip Maes, Principal Investigator — University Hospital, Antwerp; Anthe Foubert, Principal Investigator — University of Antwerp - UCLouvain; Valérie-Anne Chantrain, Principal Investigator — University of Antwerp - UCLouvain; Mira Meeus, Principal Investigator — Universiteit Antwerpen
Locations (2):
- Belgium (2):
  - University Hospital Antwerp, Edegem, Antwerp
  - Cliniques universitaires Saint-Luc, Brussels

IPD SHARING:
Plan to Share IPD: Undecided